CLINICAL TRIAL: NCT04041661
Title: The Effect of Concurrent Transcranial Direct Current Stimulation and Gait Training on Gait Performance When Doing the Cognitive Dual-task in People With Parkinson's Disease
Brief Title: Concurrent Transcranial Direct Current Stimulation and Gait Training in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19MMHIS113e
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Parkinson's Disease
Keywords: Dual task performance; Executive function; Transcrainal direct current stimulation (tDCS)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS plus gait training group (Experimental): Participants in Active tDCS plus gait training group will execute Active tDCS on left dorsolateral prefrontal cortex which combined with treadmill, 12 times per week, least 4 weeks.
  Interventions: Other: Active tDCS plus gait training
- Sham tDCS plus gait training group (Sham Comparator): Participants in Sham tDCS plus gait training group will executeSham tDCS on left dorsolateral prefrontal cortex which combined with treadmill, 12 times per week, least 4 weeks.
  Interventions: Other: Sham tDCS plus gait training

INTERVENTIONS:
Other: Active tDCS plus gait training — Participants in experimental group will accept Active tDCS which combined with treadmill
  Arms: Active tDCS plus gait training group
Other: Sham tDCS plus gait training — Participants in control group will accept Sham tDCS which combined with treadmill
  Arms: Sham tDCS plus gait training group

SUMMARY:
To investigate the effect of concurrent transcranial direct current stimulation and gait training on gait performance when doing the cognitive dual-task in people with Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic PD
* Hoehn and Yahr stages I-III
* Mini Mental Status Examination (MMSE) score ≧ 24
* Could walk 10m independently with or without gait aid

Exclusion Criteria:

* Concurrent medication likely to affect mental performance
* tDCS contraindication
* Significant neurological, vestibular, visual disorders or psychiatric illness
* Musculoskeletal or cardiopulmonary disease
* Sensory system pathology

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Dual-task walking performance | Change from baseline at 4 weeks
  To evaluate gait parameters while doing dual-task walking

SECONDARY OUTCOMES:
Single walking performance | Change from baseline at 4 weeks
  To evaluate gait parameters while doing single walking
Trail-making test A & B | Change from baseline at 4 weeks
  To evaluate executive function
Stroop color and word test-Chinese version | Change from baseline at 4 weeks
  To evaluate executive function
Digit span test | Change from baseline at 4 weeks
  To evaluate executive function